CLINICAL TRIAL: NCT03957512
Title: Heart Defects in Infants- Detection, Rescue and Care
Brief Title: Livet Skal Leves (A Life to Live)
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Holmstrøm, Professor, Oslo University Hospital
Other Study IDs: REK2010/392
Record Dates: First submitted 2019-05-18; First posted 2019-05-21 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Heart surgery — All invasive procedures

SUMMARY:
The overall objective of this project is to optimize the use of diagnostic methods and follow-up programs in infants with congenital heart defects (CHDs) in order to reduce death and complications

DETAILED DESCRIPTION:
The project is designed as retrospective cohort study based on nationwide registry data of children born 2004-16. The project group has extensive experience of similar research, and includes representatives from different fields and levels of health care.

The results will provide a solid fundament for improvement of today's clinical practice, including development of knowledge-based routines in neonatal medicine and planning of health care services. Implementation is given particular attention, and will be managed in an interdisciplinary setting. The project will be of major relevance for the patients and their families as well as medical professionals at all levels of health care.

ELIGIBILITY:
Inclusion Criteria:

* Fetuses with severe CHDs who were identified by antenatal ultrasound screening, and where the pregnancy was terminated
* Children with severe congenital heart defects born in Norway 2004-18

Exclusion Criteria:

* Lack of parental consent

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: National population
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 0-2 years
  All deaths including prenatal termination of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Holmstrøm, Dr Med, Principal Investigator — Oslo University Hospital/University of Oslo
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided